CLINICAL TRIAL: NCT03879863
Title: The RENEW Trial: A Multi-Center, Randomized, Double-Masked, Parallel-Group, Vehicle-Controlled, Adaptive Phase 3 Clinical Trial to Assess the Safety and Efficacy of Reproxalap 0.25% Ophthalmic Solution Compared to Vehicle in Subjects With Dry Eye Disease
Brief Title: The RENEW Trial: A Multi-Center, Randomized, Double-Masked, Parallel-Group, Vehicle-Controlled, Adaptive Phase 3 Clinical Trial to Assess the Safety and Efficacy of Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aldeyra Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ADX-102-DED-012
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Results first posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Reproxalap Ophthalmic Solution (0.25%) QID (Experimental)
  Interventions: Drug: Reproxalap Ophthalmic Solution (0.25%) QID
- Vehicle Ophthalmic Solution QID (Placebo Comparator)
  Interventions: Drug: Vehicle Ophthalmic Solution QID
- Reproxalap Ophthalmic Solution (0.25%) QID to BID (Experimental)
  Interventions: Drug: Reproxalap Ophthalmic Solution (0.25%) QID to BID
- Vehicle Ophthalmic Solution QID to BID (Placebo Comparator)
  Interventions: Drug: Vehicle Ophthalmic Solution QID to BID

INTERVENTIONS:
Drug: Reproxalap Ophthalmic Solution (0.25%) QID — Reproxalap Ophthalmic Solution (0.25%) administered QID for twelve weeks
  Arms: Reproxalap Ophthalmic Solution (0.25%) QID
Drug: Vehicle Ophthalmic Solution QID — Vehicle Ophthalmic Solution administered QID for twelve weeks
  Arms: Vehicle Ophthalmic Solution QID
Drug: Reproxalap Ophthalmic Solution (0.25%) QID to BID — Reproxalap Ophthalmic Solution (0.25%) administered QID for four weeks, followed by BID administration for eight weeks
  Arms: Reproxalap Ophthalmic Solution (0.25%) QID to BID
Drug: Vehicle Ophthalmic Solution QID to BID — Vehicle Ophthalmic Solution administered QID for four weeks, followed by BID administration for eight weeks
  Arms: Vehicle Ophthalmic Solution QID to BID

SUMMARY:
The RENEW Trial is a Multi-Center, Randomized, Double-Masked, Parallel-Group, Vehicle-Controlled, Adaptive Phase 3 Clinical Trial to Assess the Safety and Efficacy of Reproxalap 0.25% Ophthalmic Solution Compared to Vehicle in Subjects with Dry Eye Disease

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age of either gender and any race;
* Have a reported history of dry eye for at least 6 months prior to Visit 1;
* Have a history of use or desire to use eye drops for dry eye symptoms within 6 months of Visit 1

Exclusion Criteria:

* Have any clinically significant slit-lamp findings at Visit 1, including active blepharitis; meibomian gland dysfunction (MGD); lid margin inflammation; or active ocular allergies that require therapeutic treatment, or, in the opinion of the investigator may interfere with the assessment of the safety or efficacy of reproxalap or vehicle;
* Have or be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal) or active ocular inflammation at Visit 1;
* Have worn contact lenses within 7 days of Visit 1 or anticipate using contact lenses during the study;
* Have used any eye drops within 2 hours of Visit 1;
* Have previously had laser-assisted in situ keratomileusis (LASIK) surgery within the last 12 months;
* Have used ophthalmic cyclosporine or lifitegrast 5.0% ophthalmic solution within 90 days of Visit 1;
* Have any planned ocular and/or lid surgeries over the study period or any ocular surgery within 6 months of Visit 1;
* Have used temporary or permanent punctal plugs within 30 days prior to Visit 1 or anticipate their use during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Research Foundation, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Reproxalap Ophthalmic Solution (0.25%) QID: Reproxalap ophthalmic solution administered QID (four times daily) for twelve weeks
- Vehicle Ophthalmic Solution QID: Vehicle ophthalmic solution administered QID (four times daily) for twelve weeks
- Reproxalap Ophthalmic Solution (0.25%) QID to BID: Reproxalap ophthalmic solution administered QID (four times daily) for four weeks, followed by BID (two times daily) administration for eight weeks
- Vehicle Ophthalmic Solution QID to BID: Vehicle ophthalmic solution administered QID (four times daily) for four weeks, followed by BID (two times daily) administration for eight weeks
Period: Overall Study
Arm/Group | Reproxalap Ophthalmic Solution (0.25%) QID | Vehicle Ophthalmic Solution QID | Reproxalap Ophthalmic Solution (0.25%) QID to BID | Vehicle Ophthalmic Solution QID to BID
Started | 105 | 106 | 105 | 106
Completed | 98 | 102 | 94 | 104
Not Completed | 7 | 4 | 11 | 2

BASELINE CHARACTERISTICS:
Groups:
- Reproxalap Ophthalmic Solution (0.25%) QID: Reproxalap ophthalmic solution administered QID for twelve weeks
- Reproxalap Ophthalmic Solution (0.25%) QID to BID: Reproxalap ophthalmic solution administered QID for four weeks, followed by BID administration for eight weeks
- Total: Total of all reporting groups
Arm/Group | Reproxalap Ophthalmic Solution (0.25%) QID | Vehicle Ophthalmic Solution QID | Reproxalap Ophthalmic Solution (0.25%) QID to BID | Vehicle Ophthalmic Solution QID to BID | Total
Number analyzed (Participants) | 105 | 106 | 105 | 106 | 422
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 50 | 43 | 49 | 182
  >=65 years | 65 | 56 | 62 | 57 | 240
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 77 | 75 | 82 | 312
  Male | 27 | 29 | 30 | 24 | 110
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 8 | 8 | 33
  Not Hispanic or Latino | 96 | 98 | 97 | 98 | 389
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 0 | 0 | 3
  Asian | 4 | 4 | 8 | 9 | 25
  Black or African American | 7 | 7 | 6 | 7 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  White | 92 | 91 | 90 | 90 | 363
  Multiple | 1 | 0 | 0 | 0 | 1
  Other | 1 | 0 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 105 | 106 | 105 | 106 | 422
Iris Color (Right Eye) [Count of Participants; unit: Participants]
  Black | 1 | 1 | 0 | 1 | 3
  Blue | 32 | 38 | 34 | 26 | 130
  Brown | 41 | 37 | 44 | 53 | 175
  Hazel | 18 | 20 | 13 | 12 | 63
  Gray | 1 | 0 | 0 | 2 | 3
  Green | 12 | 10 | 14 | 12 | 48
  Other | 0 | 0 | 0 | 0 | 0
Iris Color (Left Eye) [Count of Participants; unit: Participants]
  Black | 1 | 1 | 0 | 1 | 3
  Blue | 32 | 38 | 34 | 26 | 130
  Brown | 41 | 37 | 44 | 53 | 175
  Hazel | 18 | 20 | 13 | 12 | 63
  Gray | 1 | 0 | 0 | 2 | 3
  Green | 12 | 10 | 14 | 12 | 48
  Other | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Subject-reported Ocular Dryness Score (0 - 100 Visual Analogue Scale (VAS))
Description: Change from baseline comparison of reproxalap to vehicle for subject-reported ocular dryness score VAS (0 = no discomfort - 100 = maximal discomfort), where a higher score means a worse outcome. The intervention was administered bilaterally. The least squares mean (standard error) was derived from mixed model repeated measures for change from baseline calculated using baseline score, treatment arm, visit, and the interaction of treatment arm and visit as fixed effects.
Time Frame: The efficacy assessment period (Day 1 through 85) was assessed at Weeks 1, 2, 4, 6, 8, 10, and 12; baseline was Day 1.
Population: Intent-to-treat Ocular Dryness Population with observed data only
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Reproxalap Ophthalmic Solution (0.25%) QID | Vehicle Ophthalmic Solution QID | Reproxalap Ophthalmic Solution (0.25%) QID to BID | Vehicle Ophthalmic Solution QID to BID
Number analyzed (Participants) | 85 | 86 | 85 | 85
score on a scale | -11.5 (2.44) | -15.0 (2.39) | -17.8 (2.20) | -6.8 (2.12)

2. Primary Outcome: Fluorescein Nasal Region Score (0 = None - 4 = Severe)
Description: Change from baseline comparison of reproxalap to vehicle for fluorescein staining of the nasal region (0 = none - 4 = severe), where a higher score means a worse outcome. The intervention was administered bilaterally. The least squares mean (standard error) was derived from mixed model repeated measures for change from baseline calculated using baseline fluorescein nasal score, treatment arm, visit, and the interaction of treatment arm and visit as fixed effects.
Time Frame: The efficacy assessment period (Day 15 through 85) was assessed at Weeks 2, 4, 6, 8, 10, and 12; baseline was Day 1.
Population: Intent-to-Treat Fluorescein Nasal Score Population with observed data only
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Reproxalap Ophthalmic Solution (0.25%) QID | Vehicle Ophthalmic Solution QID | Reproxalap Ophthalmic Solution (0.25%) QID to BID | Vehicle Ophthalmic Solution QID to BID
Number analyzed (Participants) | 91 | 90 | 89 | 90
units on a scale | -0.47 (0.060) | -0.46 (0.058) | -0.53 (0.056) | -0.46 (0.053)

ADVERSE EVENTS:
Time Frame: The period of time over which adverse events were collected for each subject in the clinical trial was approximately three months.
Arm/Group | Reproxalap Ophthalmic Solution (0.25%) QID | Vehicle Ophthalmic Solution QID | Reproxalap Ophthalmic Solution (0.25%) QID to BID | Vehicle Ophthalmic Solution QID to BID
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/106 | 0/105 | 0/106
Serious Adverse Events (participants affected / at risk) | 3/105 | 3/106 | 1/105 | 2/106
Other Adverse Events (participants affected / at risk) | 88/105 | 7/106 | 94/105 | 1/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Reproxalap Ophthalmic Solution (0.25%) QID (N=105) | Vehicle Ophthalmic Solution QID (N=106) | Reproxalap Ophthalmic Solution (0.25%) QID to BID (N=105) | Vehicle Ophthalmic Solution QID to BID (N=106)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 — The serious adverse event of acute kidney injury was deemed moderate in severity and not related to study drug by the Principal Investigator.
Gastroenteritis salmonella (Infections and infestations) | 1 | 0 | 0 | 0 — The serious adverse event of gastroenteritis salmonella was deemed moderate in severity and not related to study drug by the Principal Investigator.
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 — The serious adverse event of hypoxia was deemed severe in severity and not related to study drug by the Principal Investigator.
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 — The serious adverse event of pneumonia was deemed moderate in severity and not related to study drug by the Principal Investigator.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Reproxalap Ophthalmic Solution (0.25%) QID (N=105) | Vehicle Ophthalmic Solution QID (N=106) | Reproxalap Ophthalmic Solution (0.25%) QID to BID (N=105) | Vehicle Ophthalmic Solution QID to BID (N=106)
General disorders and administration site conditions (General disorders) | 88 | 7 | 94 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-03-05): https://cdn.clinicaltrials.gov/large-docs/63/NCT03879863/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/63/NCT03879863/SAP_002.pdf